CLINICAL TRIAL: NCT02865785
Title: Effect of Intralipid Infusion in Patients With Recurrent Implantation Failure (A Randomized Controlled Trial)
Brief Title: Effect of Intralipid Infusion in Patients With Recurrent Implantation Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mostafa Fouad Gomaa, Dr, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Intralipid-RIF
Record Dates: First submitted 2016-08-10; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Subfertility
Keywords: recurrent implantation failure; intralipid; uterine natural killer cells
MeSH Terms: conditions — Infertility | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Group (Active Comparator): This group will include 160 women with unexplained recurrent implantation failure undergoing a trial of IVF/ICSI. This group will receive intravenous infusion of intralipid 20% (100 mL of intralipid 20% diluted in 250 mL sterile i.v. saline administered i.v. over two hours), once between days 4 and 9 of the ovarian stimulation, and again within 7 days of a positive pregnancy test.
  Interventions: Drug: Intralipid 20%
- Placebo Group (Placebo Comparator): This group will include 160 women with unexplained recurrent implantation failure undergoing a trial of IVF/ICSI. This group will receive intravenous infusion of placebo, once between days 4 and 9 of the ovarian stimulation, and again within 7 days of a positive pregnancy test.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intralipid 20% — intralipid D4-9 of induction ovulation to be repeated within 7 days of positive pregnancy test.
  Other Names: lipofundin 20%
  Arms: Study Group
Drug: Placebo — saline infusion D4-9 of induction of ovulation to be repeated within 7 days of positive pregnancy test.
  Other Names: saline 0.9%
  Arms: Placebo Group

SUMMARY:
The aim of present study is to evaluate the effect of intralipid 20% infusion, once between days 4 and 9 of the ovarian stimulation, and again within 7 days of a positive pregnancy test on clinical pregnancy rates in women with unexplained recurrent implantation failure.

DETAILED DESCRIPTION:
The study will include 300 women with unexplained recurrent implantation failure undergoing IVF/ICSI cycle.

Randomization:

Patients fulfilling the inclusion criteria will be randomized to two groups.

Study Group:

This group will include 160 women with unexplained recurrent implantation failure undergoing a trial of IVF/ICSI. This group will receive intravenous infusion of intralipid 20%, once between days 4 and 9 of the ovarian stimulation, and again within 7 days of a positive pregnancy test.

Control Group:

This group will include 160 women with unexplained recurrent implantation failure undergoing a trial of IVF/ICSI. This group will receive intravenous infusion of placebo, once between days 4 and 9 of the ovarian stimulation, and again within 7 days of a positive pregnancy test.

Random allocation sequence generation:

A computer generated list via MedCalc ® Software, version 13.2.2 will be used, assigning each participant number to either study groups.

Allocation Concealment:

Assignment will be done by sequentially numbered, otherwise identical, sealed envelopes (SNOSE), each containing a 2-inch by 2-inch paper with a written code designating the assigned group. These papers will be placed in a folded sheet of aluminum foil fitted inside the envelope. Effort will be taken to assure absence of any detectable differences in size or weight between intervention and control envelopes. Envelopes will be chosen to be opaque and lined inside with carbon paper. Envelopes will be opened sequentially only after writing the subject's tracking information on the envelope so that the carbon paper served as an audit trail.

Blinding:

Both drug with active ingredient and placebo will be provided by the hospital pharmacy in identical sealed opaque containers, equal in weight, similar in appearance, and tamper-proof. The drug with the active ingredient containers will be labeled either Group A or Group B by the head pharmacist and the assignment kept secret to be revealed after the end of the study.

Drugs will be administered to patients by a sealed opaque infusion drip.

An endometrial biopsy (Wallach endocell sampler ® ) will be taken during the luteal phase of the menstrual cycle and put in formalin. The biopsy will be embedded in paraffin, cut into sections and immunohistochemistry will be used to identify uNK cells using an antibody to CD56 and CD16 (NCL-CD56-16; Novacastra ® ). A cut-off of normality of 5% uNK cell density will be used.

IVF/ICSI cycle will be done using the standard LLP in both groups.

primary outcome will be Live birth rate.

secondary outcomes will be biochemical and clinical pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-38 years of age.
2. Recurrent implantation failure, defined as failure to achieve a recognizable intrauterine gestational sac by ultrasonography after transfer of at least four good-quality embryos in a minimum of three fresh or frozen IVF cycles (Coughlan et al, 2014).

   Good-quality embryos will be defined as those characterized by absence of multinucleated blastomeres, four or five blastomeres on day 2, seven or more cells on day 3, and ≤ 20% anucleated fragments (Van Royen et al, 1999).
3. Normal transvaginal ultrasonography
4. Normal office hysteroscopy.
5. Normal hysterosalpingography.
6. Absence of any structural pathological findings in laparoscopy.
7. Normal male and female karyotyping.
8. Normal endocrinological profile during ovarian stimulation
9. Normal anti-cardiolipin antibody IgG, IgM and lupus anticoagulant.
10. Normal thrombophilia screen in the form of protein C, protein S, anti thrombin III, factor V mutations and factor V leiden.
11. Elevated uterine natural killer cells (uNK) density in luteal phase endometrial biopsy, defined as ≥ 5% CD16+ CD56+ cells in the stroma underlying the luminal epithelium (Tang et al, 2013; Quenby et al, 2005).
12. Normal parameters of male semen analysis according to WHO criteria 2010.
13. Written and signed informed consent by the patient to participate in the study.

Exclusion Criteria:

1. Age more than 38 years.
2. Less than 3 failed IVF cycles.
3. Poor embryo quality in previous IVF trials.
4. Abnormal ultrasonographic finding, e.g. endometrial polyps, fibroids or ovarian cysts.
5. Abnormal hysteroscopic finding, e.g. endometrial polyps, endometrial hyperplasia or fibroid.
6. Abnormal hysterosalpingographic finding, e.g. hydrosalpinx or peritoneal adhesions.
7. Abnormal male or female karyotyping.
8. Abnormal endocrinological profile during ovarian stimulation, e.g. hyperprolactinemia
9. Expected poor ovarian responders according to Bologna criteria (Ferraretti et al, 2011), i.e. presence of at least two of the following three features:

   * Presence of risk factor for poor ovarian response (POR) represented by advanced maternal age (≥ 40 years) or any other genetic or acquired conditions possibly linked to a reduced amount of resting follicles.
   * A previous POR, represented by a cycle cancelled (following the development of less than three growing follicles) or the collection of less than four oocytes in response to an ovarian stimulation protocol of at least 150 IU FSH per day.
   * An abnormal ovarian reserve test (i.e. AFC < 5-7 follicles or AMH < 0.5-1.1 ng/ml).
10. Positive anticardiolipin antibodies or lupus anticoagulant.
11. Positive thrombophilia screen.
12. Normal uterine natural killer cells (uNK) density in luteal phase endometrial biopsy, defined as < 5% CD16+ CD56+ cells in the stroma underlying the luminal epithelium (Tang et al, 2013; Quenby et al, 2005).
13. Abnormal semen analysis parameters according to WHO criteria 2010.
14. Any chronic medical disorder, e.g. hypertension, autoimmune disorders, … etc.
15. Known allergy to any of the intralipid constituents.
16. Mental condition rendering the patients unable to understand the nature, scope and possible consequences of the study.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 38 gestational weeks

SECONDARY OUTCOMES:
Clinical pregnancy rate | 6 gestational weeks
Chemical pregnancy rate | 6 gestational weeks

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Afifi, MBBCH, Study Director — Resident of O&G
Locations (1):
- AinShams Maternity Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No